CLINICAL TRIAL: NCT07397754
Title: Sodium-rich COndiments Unifying Health and Taste
Acronym: Scout
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Darel Toh, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2025-063
Record Dates: First submitted 2025-11-18; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Elevated Blood Pressure; Vascular Health; Sensory Evaluation
Keywords: sodium intake; natremic index; elevated blood pressure; cardiometabolic outcomes; condiments; Asian; vascular health; sensory evaluation
MeSH Terms: conditions — Hypertension | interventions — Sodium Chloride, Dietary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control porridge with no condiments (Experimental): This arm will consist of plain porridge which participants will consume.
  Interventions: Other: Control porridge with no condiments
- Porridge with light soya sauce (Experimental): This arm will consist of plain porridge with light soya sauce which participants will consume.
  Interventions: Other: Porridge with light soya sauce
- Porridge with fermented bean paste (Experimental): This arm will consist of plain porridge with fermented bean paste which participants will consume.
  Interventions: Other: Porridge with fermented bean paste
- Porridge with table salt (Experimental): This arm will consist of plain porridge with table salt which participants will consume.
  Interventions: Other: Porridge with table salt

INTERVENTIONS:
Other: Control porridge with no condiments — To examine acute cardiovascular health response to plain porridge.
  Arms: Control porridge with no condiments
Other: Porridge with light soya sauce — To examine acute cardiovascular health response to plain porridge with saltiness-matched light soya sauce
  Arms: Porridge with light soya sauce
Other: Porridge with fermented bean paste — To examine acute cardiovascular health response to plain porridge with saltiness-matched fermented bean paste
  Arms: Porridge with fermented bean paste
Other: Porridge with table salt — To examine acute cardiovascular health response to plain porridge with saltiness-matched table salt.
  Arms: Porridge with table salt

SUMMARY:
This research aims to develop an evidence-based classification for sodium-rich condiments (natremic index) based on their CVD-related risks. It is hypothesised that the acute cardiovascular and physiological response (effectively extrapolated to long-term CVD risks) to meals prepared with various sodium-rich condiments can be leveraged upon for the development of such an index that will systematically classify sodium-rich condiments based on the risk they present to cardiovascular health.

DETAILED DESCRIPTION:
Hypertension is the leading risk factor for cardiovascular diseases (CVDs) in older adults. While absolute dietary sodium reductions remain vital for prevention, effective long-term management must take stock of sensorial efficacy and acceptance, alongside the corresponding impacts on health. In Asia, this phenomenon is distinct due to a genetic predisposition of the population to salt sensitivity (increased risk), and a distinct food culture characterised by regional condiments (e.g. soy sauce, fermented bean paste).

The aim of this research is to develop an evidence-based classification for sodium-rich condiments (natremic index) based on their CVD-related risks. Perceived saltiness intensity is influenced by factors beyond the total amount of sodium consumed (e.g. flavour enhancers like MSG, tastes synergism etc.).

Similarly, while hypertension is predisposed by excessive sodium intake, growing evidence also suggests the potential role of bioactive compounds and ingredients (including some identified from Asian-style condiments e.g. spices, soya-derived flavonoids) that may elicit cardiovascular protective properties.

Contrary to generic recommendations that focused solely on absolute sodium reduction, sustainable solutions must simultaneously address concerns surrounding long-term health and consumer acceptance.

Much like the well-established glycemic index, it is hypothesised that the development of a natremic index, designed to evaluate and classify sodium-rich condiments according to their risks to cardiovascular health will serve as a vital, first of its kind strategy that can reliably guide public health recommendations, and spearhead next-generation innovations in the food and nutrition industry. The proposed research is split into two main parts that will investigate in detail three sodium-rich condiments commonly used in Asia cuisines: light soy sauce (condiment 1), fermented bean paste (condiment 2), and table salt (control), from sensory and health perspectives

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 50, < 75 years old
2. Male or postmenopausal female (self-reported)
3. ≥ 50 kg body weight
4. Systolic blood pressure (≥ 130, < 160 mmHg) or diastolic blood pressure (≥ 85, < 100 mmHg)
5. Willing and able to follow intervention protocol
6. Ability to identify basic tastes (determined by taste discrimination test)
7. English speaking

Exclusion Criteria:

1. Prescribed and taking medication which may affect study outcomes (i.e. for blood pressure management, blood thinning etc.) in consultation with study physician (Prof Melvin Leow) and PI(Dr Darel Toh)
2. Type 1 or type 2 diabetes mellitus (i.e. fasting blood glucose ≥ 7.0 mmol/L or HbA1c ≥ 6.5 %)
3. Taking dietary supplements which may affect study outcomes one month prior to their first visit in consultation with study physician, PI and study team
4. Obesity (BMI ≥ 27.5 kg/m2)
5. History or known present diagnosis of hematological (G6PD and coagulation disorders), hepatic (hepatitis B and C), renal, gastrointestional or other relevant disease / disorders which may affect the outcomes of interest in consultation with study physician, PI and study team
6. History of arteriovenous shunt or mastectomy
7. Women who are pregnant, lactating or planning pregnancy
8. History or present diagnosis of HIV and/or tuberculosis
9. History of severe vasovagal syncope (blackouts or near faints) following blood draw
10. Drug abuse within last 5 years
11. Excessive alcoholic beverage consumption > 2 servings per day (1 serving defined as 360 mL beer, 150 mL wine or 45 mL distilled spirits)
12. Smoking (cigarette, e-cigarette, cigar, pipe, vape)
13. Engaging in habitual vigorous physical activity (as defined by physical activity questionnaire-PAR)
14. Allergic or intolerance to intervention foods.
15. Dislike or unwilling to consume intervention foods
16. Photophobic (sensitivity to intense lights and colours), particularly to intense red lights
17. Has sinus problems problems that affect taste and smell
18. Involvement in other clinical studies that may influence the outcome of the study
19. An ASTAR Staff.
20. A study team member or their immediate family member

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Endopat assessment | EndoPAT assessments which will serve as the primary outcome of interest will be measured at postprandial intervals (up to 3 measurements) over 4 hours.
  EndoPAT test which will measure endothelial health and function at baseline. The EndoPAT test is a non-invasive procedure that involves the placement of probes on each index finger, followed by blood pressure cuff inflation for measurements of the arterial tone and blood flow responses (e.g. EndoPAT index).

SECONDARY OUTCOMES:
Ambulatory blood pressure | 24 hour period consisting of: Postprandially 15 minutes intervals (over 4 hours), 30 minutes interval (after 4 hours)
  The ambulatory blood pressure monitor will be attached and programmed for blood pressure measurements at pre-determined intervals. Blood pressure measurements will be taken at 15 minutes interval during the postprandial study duration (4 hours), 30 minutes interval (after the 4 hours) when participant is awake, and hourly when the participants are asleep. During each measurement, participants must be standing, seated or lie still, stay relaxed and silent. If seated they should keep their feet flat on the floor (not crossed).
Palatability questionnaire rated on a visual analogue scale "Good" to "Bad" | Test meal is consumed for 15 minutes. At the end of 15 minutes, palatibility questionnaire is completed.
  Palatability appetite questionnaire, rated on a visual analogue scale. To place a vertical mark on the thick line to indicate how person feels at that moment in response to various questions. At opposite ends of each line are descriptors which should be read carefully before placing the vertical line.
Serum and Plasma sodium and potassium | Blood will be sampled at timepoints, t = 0 minute (Baseline) and at t = 30, 45, 60, 120, 180, 240 minute for each session
  Serum and plasma collected are for sodium and potassium assessment
Subjective appetite questionnaire | t=0 minute (Baseline), and t= 30, 45, 60, 120, 180, 240 minute for each session.
  Subjective appetite questionnaire, rated on a 0-100 visual analogue scale. 0 corresponds to "not at all" and 100 corresponds to "extremely".Questions usually used are "How hungry are you?" "How full are you?" "How strong is your desire to eat?" "How much food do you think you could eat?"
Taste acuity test | Test administered once at each session (5 sessions). Each test takes 20 minutes.
  Sensory method to assess participant's recognition, detection and aversion threshold for sweet, salty, umami, sour and bitter taste. Up to 25 samples (approximately 10 milimetre each) will be evaluated per test session.
Ultrasound scan of carotid intima-media thickness | At baseline only
  The ultrasound scan measures the thickness of the carotid intima-media layers on the side of the neck which is a marker for CVD risk
Evaluation | Administered during session4, 5 and 6. Each evaluation takes1 hour.There is a 1-minute inter-stimulus break between each sample for palate cleansing.
  Participants will taste up to 25 test samples (undosed or dosed with various condiments with varying concentrations). A mandatory inter-stimulus break of one-minute is enforced between each sample to reduce possible fatigue and allow time for palate cleansing. The QDA method features participants rating pre-defined sensory attributes (e.g. salty taste intensity) on a 0-100 VAS scale. During sample evaluation, participants will be instructed to place the entire sample in their mouth, hold it in, swirl for 5 seconds before swallowing, then rate the taste intensity of the sample marked from 'low' (0) to 'high' (100) on a scale in Compusense

OTHER OUTCOMES:
Health and lifestyle relevant questionnaire to to assess eligibility for inclusion/exclusion criteria. | This is conducted at the Screening Visit, 1 time only. Takes 15 minutes to complete.
  This is to evaluate the participants eligibility for the study. Section A: Participant information, Section B: Medical and Health History, Section C: Lifestyle and Diet. Section A, B and C are questions with "Yes" or "No" to be answered. Section D: Physical Acitvity where participants select only one description that best represents their usual physical activity for leisure over the past 3 months.
3 day food records | Administered once during whole study. Record 3 days of food intake (over 72 hours). Recording can range from 5-15 minutes for every meal recorded (recording duration depends on how many meals to be recorded for the day)
  Dietary intake will be assessed by documenting all foods and beverages consumed over 3 consecutive days, typically including 2 weekdays and 1 weekend day. Participants will record all foods and beverages consumed using household measures.
Gastrointestinal Symptom Rating Scale (GSRS) | Administered once over the course of the study. Takes about 1-2 minutes to complete each item.
  The Gastrointestinal Symptom Rating Scale (GSRS) is a validated, self-administered questionnaire used to assess the severity of gastrointestinal symptoms. It consists of 15 items grouped into five symptom domains: reflux, abdominal pain, indigestion, diarrhoea, and constipation. Each item is rated on a 7-point Likert scale ranging from 1 (no discomfort) to 7 (very severe discomfort). Higher scores indicate greater gastrointestinal symptom severity.
Council on Nutrition Appetite Questionnaire (CNAQ)- Rate items like appetite quality, fullness, hunger, taste of food, and eating frequency on a 5-point Likert scale (e.g., from "very poor" to "very good"). A total score is often used. | Administered only once over the course of the study. Takes about 1-2 minutes to complete each item.
  An 8-item self-reported appetite assessment tool used in clinical research to evaluate appetite status.
Pittsburgh Sleep Quality Index (PSQI)- Self-rated items,combined to generate 7 component scores to obtain a global PSQI score ranging from 0 to 21, with higher scores indicating poorer sleep quality | Administered only once over the course of the study. Takes about 1-2 minutes to complete each item
  Validated, self-administered questionnaire used to assess subjective sleep quality and sleep disturbances over the previous 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No